CLINICAL TRIAL: NCT00670501
Title: Effects of LY333334 in the Treatment of Postmenopausal Women With Osteoporosis
Brief Title: Effects of Teriparatide in the Treatment of Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 547; B3D-MC-GHAC
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): LY333334 40 micrograms/day plus calcium and vitamin D
  Interventions: Drug: teriparatide; Drug: Calcium Supplement; Drug: Vitamin D Supplement
- 2 (Experimental): LY333334 20 micrograms/day plus calcium and vitamin D
  Interventions: Drug: teriparatide; Drug: Calcium Supplement; Drug: Vitamin D Supplement
- 3 (Placebo Comparator): Placebo plus calcium and vitamin D
  Interventions: Drug: Placebo; Drug: Calcium Supplement; Drug: Vitamin D Supplement

INTERVENTIONS:
Drug: teriparatide — 40 micrograms/day subcutaneous injection for 3 years with optional 2 year extension phase
  Other Names: LY333334; Forteo; Forsteo
  Arms: 1
Drug: teriparatide — 20 micrograms/day subcutaneous injection for 3 years with optional 2 year extension phase
  Other Names: LY333334; Forteo; Forsteo
  Arms: 2
Drug: Placebo — Placebo for subcutaneous injection will be supplied in a prefilled injection device with a cartridge identical in appearance to the LY333334 device.
  Arms: 3
Drug: Calcium Supplement — Approximately 1000 mg/day of elemental calcium will be supplied as open-label oral supplement
Drug: Vitamin D Supplement — Approximately 400 to 1200 IU/day of vitamin D will be supplied as open-label oral supplement

SUMMARY:
The primary objective of this study is to demonstrate a reduction in the proportion of new vertebral fractures in postmenopausal women with osteoporosis following 3-years of treatment with 20 and 40 mcg/day of teriparatide plus calcium and vitamin D compared with calcium and vitamin D alone.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women.
* A minimum of either one moderate or two mild atraumatic vertebral fractures, and a minimum of seven evaluable nonfractured vertebrae.
* Hip BMD or lumbar spine BMD measurement at least 1.0 standard deviation (SD) below the average bone mass for young, healthy women (T-score) only in patients with fewer than two moderate fractures or in patients previously treated with therapeutic doses of bisphosphonates or fluorides
* Normal or clinically nonsignificant abnormal laboratory values (serum calcium, PTH(1-84), & urine calcium must be within normal limits at baseline; 25-hydroxyvitamin D must be between the lower limit of normal & 3 times the upper limit of normal at baseline).

Exclusion Criteria:

* Fractures in areas of bone affected by diseases other than osteoporosis (for example, cancer or Paget's disease).
* Satisfactory baseline thoracic and lumbar spinal x-ray views cannot be obtained as determined by the centralized x-ray quality assurance center (for example, severe scoliosis or kyphosis).
* Current or recent (within 1 year prior to randomization) metabolic bone disorders other than postmenopausal osteoporosis, such as Paget's disease, renal osteodystrophy, osteomalacia, or any secondary causes of osteoporosis
* Current or recent (within 1 year prior to randomization) disease which affects bone metabolism, such as hypoparathyroidism, hyperparathyroidism, or hyperthyroidism.
* Currently suspected carcinoma or history of carcinoma in the 5 years prior to randomization.
* Nephrolithiasis or urolithiasis in the 2 years prior to randomization.
* Current or recent (within 1 year prior to randomization) sprue, inflammatory bowel disease, or malabsorption syndrome, or any indication of poor intestinal absorption of calcium, such as the combination of a low urinary calcium excretion and an elevated serum intact parathyroid hormone level.
* Poor medical or psychiatric risk for treatment with an investigational drug, in the opinion of the investigator.
* Treatment with androgens or other anabolic steroids in the 6 months prior to randomization.
* Treatment with calcitonins in the 2 months prior to randomization.
* Treatment with estrogen
* Treatment with progestins in the 3 calendar months prior to randomization, or for more than 2 months in the 12 calendar months prior to randomization.
* Treatment with corticosteroids.
* Treatment with fluorides in the 6 months prior to randomization or for more than 60 days in the 24 months prior to randomization.
* Treatment with oral bisphosphonates in the 3 months prior to randomization or for more than 60 days in the 24 months prior to randomization; treatment with intravenous bisphosphonates in the 24 months prior to randomization.
* Treatment with vitamin D >50,000 IU/week, or with any dose of calcitriol, analogs, or agonists in the 6 months prior to randomization. The 25-hydroxyvitamin D laboratory value at randomization must be between the lower limit of normal and three times the upper limit of normal.
* Treatment with coumarins and indandione derivatives in the 3 months prior to randomization; treatment with heparins >10,000 U/day for more than 30 days in the 6 months prior to randomization.
* Treatment with calcium- or aluminum-containing antacids
* Treatment with any other drug known to affect bone metabolism in the 6 months prior to randomization.
* Treatment with any investigational drug during the month prior to the calcium and vitamin D run-in phase. Treatment with investigational drugs in certain therapeutic classes during the month prior to the calcium & vitamin D run-in phase.

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1637 (Actual)
Dates: Start 1996-08; Primary Completion 1999-04 (Actual); Study Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate a reduction in the proportion of patients with new vertebral fractures (by spinal x-ray) following 3-year treatment with 20 and 40 micrograms/day of LY333334 plus calcium and vitamin D compared with calcium and vitamin D alone. | Baseline, randomization, 24 , 36, and 60 months

SECONDARY OUTCOMES:
To establish the effect of long-term treatment with LY333334 plus calcium and vitamin D, compared with calcium and vitamin D alone, on lumbar spine and hip BMD in postmenopausal women with osteoporosis | Lumbar Spine: Randomization -2wks, Randomization,( 3 & 6 months in a subset of pts), 12 , 18 , 24 , 36 , 48 & 60 months. Hip BMD: Randomization -2wks, Randomization, 12 , 24 , 36 , 48 & 60 months.
To establish the effect of long-term treatment with LY333334 plus calcium and vitamin D, compared with calcium and vitamin D alone, on total body and radial (forearm) BMD in postmenopausal women with osteoporosis at selected study sites | Randomization, 12, 24, 36, 48 and 60 months
To establish the effect of long-term treatment with LY333334 plus calcium and vitamin D, compared with calcium and vitamin D alone, on the rate of new vertebral fractures (by spinal x-ray) in postmenopausal women with osteoporosis. | Baseline, randomization, 24 months, 60 months
To establish the effect of treatment with LY333334 plus calcium & vitamin D, compared with calcium & vitamin D alone, by x-ray on the proportion of subjects experiencing new nonvertebral fractures alone & new nonvertebral & vertebral fractures combined. | As clinically needed throughout the trial
To assess the effect of long-term treatment with LY333334 plus calcium and vitamin D, compared with calcium and vitamin D alone, on height (via Harpenden stadiometer or other suitable stadiometer) in postmenopausal women with osteoporosis | Randomization, 12, 24, 36, 48, and 60 months
To determine the histomorphometric effects of LY333334 plus calcium & vitamin D, compared with calcium & vitamin D alone by biopsy, on the iliac crest (bone formation & resorption, mineralization, and trabecular structure) in a subset of subjects. | Randomization, 12 and 24 months
To assess effects of LY333334 plus calcium & vitamin D, compared with calcium & vitamin D alone, on biochemical markers of bone formation & resorption (bone-specific alkaline phosphatase, PICP, urinary N-telopeptide, & urinary free deoxypyridinolines) | Randomization, 1, 3, 6, 12, 24, 36, 48, and 60 months
To assess population pharmacokinetics of LY333334 at selected study sites. Nonlinear mixed effect modeling [NONMEM])and or PTH(1-84) will be employed to evaluate serum concentrations of LY333334. | Months 1, 3, 6, 12, 18, 24, 30, 36 and 60
To quantify medical resources used by patients during the study so that a cost-effectiveness analysis can be performed. | Randomization, 6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 Months
To assess the impact of LY333334 on health-related quality of life in postmenopausal women with osteoporosis. Quality of life instruments will be completed where translated and validated instruments are available. | Randomization, 12, 24, 36, 48, and 60 months
To establish the safety of chronic administration of LY333334 in postmenopausal women with osteoporosis. Adverse events, physical examinations and laboratory tests will be used to assess safety in the patients. | Adverse Events: throughout the trial. Labs:Baseline, randomization, 1, 6, 12, 24, 36, 48, and 60 months. Physical Exams: 12, 24, 36, 48, and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CT LILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Capital Federal, Argentina
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels, Belgium
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague, Czechia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus, Denmark
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio, Finland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged, Hungary
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky, Israel
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arenzano, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam, Netherlands
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch, New Zealand
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kristiansand, Norway
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw, Poland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala, Sweden

REFERENCES:
- [Derived] Prevrhal S, Krege JH, Chen P, Genant H, Black DM. Teriparatide vertebral fracture risk reduction determined by quantitative and qualitative radiographic assessment. Curr Med Res Opin. 2009 Apr;25(4):921-8. doi: 10.1185/03007990902790993. PMID 19250060